CLINICAL TRIAL: NCT02752958
Title: Study to Investigate the Impact on Oral Health Related Quality of Life of Managing Dentine Hypersensitivity With a Daily Use Anti-Sensitivity Toothpaste
Brief Title: Impact of Long Term Management of Dentine Hypersensitivity (DH) With a Daily Use Anti-sensitivity Toothpaste on the Quality of Life Related to Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 204930
Record Dates: First submitted 2016-04-25; First posted 2016-04-27 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-06

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tin Fluorides

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- stannous fluoride (Experimental): This was a non-comparative design study, all the participants applied dentifrice containing stannous fluoride for 1 timed minute, twice daily (morning and evening) for 24 weeks.
  Interventions: Drug: stannous fluoride

INTERVENTIONS:
Drug: stannous fluoride — 0.454% w/w (weight per weight) stannous fluoride

SUMMARY:
This multicentre, non-comparative design study will monitor the impact of long term management of DH with daily use of a sensitivity toothpaste on the quality of life of a population of sensitivity sufferers. Changes in oral health related quality of life will be monitored using the Dentine Hypersensitivity Experience Questionnaire (DHEQ). The study will be conducted in participants in good general health, with pre-existing self-reported and clinically diagnosed tooth sensitivity at screening.

DETAILED DESCRIPTION:
This will be multicenter, non-comparative design to monitor the impact of long term management of DH with daily use of a sensitivity toothpaste on the quality of life of a population of sensitivity sufferers, using the DHEQ. Changes in DH will be monitored clinically over the 24 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy ofthe informed consent form
* Aged 18-55 years
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: No clinically significant and relevant abnormalities of medical history or oral examination and absence of any condition that would impact on the participant's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements
* Understands and is willing, able and likely to comply with all study procedures and restrictions
* At Visit 1 (Screening): Self-reported his of dentinal hypersensitivity (DH) lasting more than six months but not more than 10 years, minimum of 20 natural teeth, Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, that meet all of the following criteria: Signs of facial/cervical gingival recession and/or signs of erosion or abrasion (EAR).Tooth with MGI score =0 adjacent to the test area (exposed dentine) only [Lobene, 1986] and a clinical mobility of ≤1 Tooth with signs of sensitivity measured by qualifying evaporative air assessment (Y/N response)
* At Visit 2 (Baseline): Minimum of two, non-adjacent accessible teeth (incisors, canines, premolars), that meet all of the following criteria: with signs of sensitivity, measured by a qualifying evaporative air assessment (Schiff Sensitivity Score ≥ 2)

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study
* Women who are breast-feeding
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit.

and previous participation in this study

* Recent history (within the last year) of alcohol or other substance abuse
* An employee of the sponsor or the study site or members of their immediate family
* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes and any condition which, in the opinion of the investigator, causes xerostomia
* Dental prophylaxis within 4 weeks of Screening, tongue or lip piercing or presence of dental implants, desensitizing treatment within 8 weeks of Screening (professional sensitivity, treatments and non-dentifrice sensitivity treatments), gross periodontal disease, treatment of periodontal disease (including surgery)within 12 months of Screening, scaling or root planning within 3 months of Screening and teeth bleaching within 8 weeks of Screening
* Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of Screening, tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine and Sensitive tooth not expected to respond to treatment with an over-the-counter dentifrice in the opinion of the investigator
* Use of an oral care product indicated for the relief of dentine hypersensitivity within 8 weeks of screening (participants will be required to bring their current oral care products to the site in order to verify the absence of known anti-sensitivity ingredients)
* Daily doses of medication/treatments which, in the opinion of the investigator, could interfere with the perception of pain. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilizers, anti-depressants, mood-altering and anti-inflammatory drugs, currently taking antibiotics or has taken antibiotics within 2 weeks of Baseline and daily dose of a medication which, in the opinion of the investigator, is causing xerostomia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Ellesmere Port, Cheshire
  - GSK Investigational Site, Widnes, Cheshire

REFERENCES:
- [Derived] Mason S, Burnett GR, Patel N, Patil A, Maclure R. Impact of toothpaste on oral health-related quality of life in people with dentine hypersensitivity. BMC Oral Health. 2019 Oct 22;19(1):226. doi: 10.1186/s12903-019-0919-x. PMID 31640741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had 2 centers in United Kingdom (UK) but, all the participants were recruited from the 1 center only.
Pre-assignment Details: A total of 163 participants were screened, of which 75 participants were enrolled and randomized in the study. A total of 88 participants were not randomized in study as 53 participants did not meet study criteria, 1 participant had adverse event (AE), 3 were lost to follow up, 6 had protocol violation and 25 due to other reason (not specified).
Groups:
- Overall Study: Stannous Fluoride: This was a non-comparative design study, all the participants applied dentifrice containing 0.454% weight by weight (w/w) stannous fluoride for 1 timed minute, twice daily (morning and evening) for 24 weeks.
Period: Overall Study
Arm/Group | Overall Study: Stannous Fluoride
Started | 75
Completed | 66
Not Completed | 9
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2
Not completed — Other (Reason not specified) | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were randomised and received at least 1 dose of study treatment.
Groups:
- Stannous Fluoride: Participants applied dentifrice containing 0.454% w/w stannous fluoride for 1 timed minute, twice daily (morning and evening).
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.2 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 75
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Total Score (34 Item Total From Section 2) of Dentine Hyersensitivity Experience Questionnaire (DHEQ) at Week 4
Description: All participants scored first 34 questions present in section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6=Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Section 2 had questions about the ways in which the sensations in the teeth affected participants in daily life. It was grouped into domains as follows: Restrictions (Section 2, Q1-4), Adaptation (Section 2, Q5-16), Social Impact (Section 2, Q17 to 21), Emotional Impact (Section 2, Q22 to 29), and Identity (Section 2, Q30 to 34).
Time Frame: At Baseline and Week 4
Population: The intention to treat (ITT) population was the primary population of analysis, defined as all participants who received the study toothpaste and had at least one post - baseline DHEQ/clinical assessment.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Stannous Fluoride: All the participants applied dentifrice containing 0.454% w/w stannous fluoride for 1 timed minute, twice daily (morning and evening) for 24 weeks.
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a Scale
  At Baseline | 142.41 (36.084)
  At Week 4: number analyzed (Participants) | 67
  At Week 4 | 135.24 (34.745)
  Change from Baseline at Week 4: number analyzed (Participants) | 67
  Change from Baseline at Week 4 | -6.28 (22.852)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 (Baseline ) versus (vs.) Week 4; Test type: Other; p = 0.0944, ANOVA; From ANOVA model with visit and site as fixed effect and subject as random effect. Visit*site interaction included where significant at 10% level; Mean Difference (Final Values) = 5.89, 95% CI 2-sided [-1.018 to 12.80] — Difference is the baseline score minus Week 4 score such that a positive difference favour to test dentifrice. Week 0 = Baseline Value

2. Primary Outcome: Change From Baseline in Mean Total Score (34 Item Total From Section 2) of Dentine Hyersensitivity Experience Questionnaire (DHEQ) at Week 8
Description: as for outcome 1
Time Frame: At Baseline and Week 8
Population: ITT population was the primary population of analysis, defined as all participants who received the study toothpaste and had at least one post - baseline DHEQ/clinical assessment.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a Scale
  At Baseline | 142.41 (36.084)
  At Week 8: number analyzed (Participants) | 69
  At Week 8 | 126.58 (42.131)
  Change from Baseline at Week 8: number analyzed (Participants) | 69
  Change from Baseline at Week 8 | -16.33 (32.512)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 (baseline) vs. Week 8; Test type: Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 16.99, 95% CI 2-sided [10.128 to 23.849] — Difference is the baseline score minus other weeks score such that a positive difference favour to test dentifrice. Week 0 = Baseline Value

3. Primary Outcome: Change From Baseline in Mean Total Score (34 Item Total From Section 2) of Dentine Hyersensitivity Experience Questionnaire (DHEQ) at Week 12
Description: as for outcome 1
Time Frame: At Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score ona Scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score ona Scale
  At Baseline | 142.41 (36.084)
  At Week 12: number analyzed (Participants) | 70
  At Week 12 | 120.39 (44.694)
  Change from Baseline at Week 12: number analyzed (Participants) | 70
  Change from Baseline at Week 12 | -22.54 (39.724)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 (baseline) vs. Week 12; Test type: Other; p < 0.0001, ANOVA; From ANOVA model with visit and site as fixed effect and participant as random effect. Visit*site interaction included where significant at 10% level; Mean Difference (Final Values) = 22.70, 95% CI 2-sided [15.870 to 29.539] — [estimate comment as in outcome 2, analysis 1]

4. Primary Outcome: Change From Baseline in Mean Total Score (34 Item Total From Section 2) of Dentine Hyersensitivity Experience Questionnaire (DHEQ) at Week 16
Description: All participants scored first 34 questions present in section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6=Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Section 2 had questions about the ways in which the sensations in the teeth affect participants in daily life. It was grouped into domains as follows: Restrictions (Section 2, Q1-4), Adaptation (Section 2, Q5-16), Social Impact (Section 2, Q17 to 21), Emotional Impact (Section 2, Q22 to 29), and Identity (Section 2, Q30 to 34).
Time Frame: At Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score ona Scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score ona Scale
  At Baseline | 142.41 (36.084)
  At Week 16: number analyzed (Participants) | 66
  At Week 16 | 115.36 (43.977)
  Change from Baseline at Week 16: number analyzed (Participants) | 66
  Change from Baseline at Week 16 | -27.68 (38.654)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 (baseline) vs. Week 16; Test type: Other; p < 0.0001, ANOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 27.21, 95% CI 2-sided [20.245 to 34.165] — [estimate comment as in outcome 2, analysis 1]

5. Primary Outcome: Change From Baseline in Mean Total Score (34 Item Total From Section 2) of Dentine Hyersensitivity Experience Questionnaire (DHEQ) at Week 20
Description: as for outcome 4
Time Frame: At Baseline and Week 20
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a Scale
  At Baseline | 142.41 (36.084)
  At Week 20: number analyzed (Participants) | 66
  At Week 20 | 112.32 (49.163)
  Change from Baseline at Week 20: number analyzed (Participants) | 66
  Change from Baseline at Week 20 | -30.58 (42.591)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 20; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 31.42, 95% CI 2-sided [24.464 to 38.385]

6. Primary Outcome: Change From Baseline in Mean Total Score (34 Item Total From Section 2) of Dentine Hyersensitivity Experience Questionnaire (DHEQ) at Week 24
Description: as for outcome 1
Time Frame: At Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a Scale
  At Baseline | 142.41 (36.084)
  At Week 24: number analyzed (Participants) | 66
  At Week 24 | 111.20 (50.179)
  Change from Baseline at Week 24: number analyzed (Participants) | 66
  Change from Baseline at Week 24 | -31.70 (44.268)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 (baseline) vs. Week 24; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 32.55, 95% CI 2-sided [25.585 to 39.506] — [estimate comment as in outcome 2, analysis 1]

7. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Restrictions (4 Item Total From Section 2 Questions 1 to 4) at Week 4
Description: All participants scored first 4 questions present in Domain Restriction of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6=Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Restriction domain consisted of following questions Q1: Having sensation in my teeth takes a lot of the pleasure out of eating and drinking, Q2: there have been times when I can't finish my meal because of the sensations, Q3: It takes a long time to finish some foods and drinks because of sensations, and Q4: there have been times when I have had problems eating ice cream because if these sensations.
Time Frame: At Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 19.55 (5.088)
  At Week 4: number analyzed (Participants) | 67
  At Week 4 | 18.24 (4.707)
  Change from Baseline at Week 4: number analyzed (Participants) | 67
  Change from Baseline at Week 4 | -1.21 (4.021)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs. Week 4; Test type: Other; p = 0.0312, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.18, 95% CI 2-sided [0.108 to 2.262] — [estimate comment as in outcome 2, analysis 1]

8. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Restrictions (4 Item Total From Section 2 Questions 1 to 4) at Week 8
Description: as for outcome 7
Time Frame: At Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score ona scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score ona scale
  At Baseline | 19.55 (5.088)
  At Week 8: number analyzed (Participants) | 69
  At Week 8 | 16.86 (5.712)
  Change from Baseline at Week 8: number analyzed (Participants) | 69
  Change from Baseline at Week 8 | -2.75 (4.924)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 8; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.80, 95% CI 2-sided [1.728 to 3.866] — [estimate comment as in outcome 2, analysis 1]

9. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Restrictions (4 Item Total From Section 2 Questions 1 to 4) at Week 12
Description: as for outcome 7
Time Frame: At Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 19.55 (5.088)
  At Week 12: number analyzed (Participants) | 70
  At Week 12 | 16.31 (6.147)
  Change from Baseline at Week 12: number analyzed (Participants) | 70
  Change from Baseline at Week 12 | -3.19 (5.619)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs. Week 12; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.26, 95% CI 2-sided [2.192 to 4.322] — [estimate comment as in outcome 2, analysis 1]

10. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Restrictions (4 Item Total From Section 2 Questions 1 to 4) at Week 16
Description: as for outcome 7
Time Frame: At Baseline and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a Scale
  At Baseline | 19.55 (5.088)
  At Week 16: number analyzed (Participants) | 66
  At Week 16 | 15.55 (5.786)
  Change from Baseline at Week 16: number analyzed (Participants) | 66
  Change from Baseline at Week 16 | -3.98 (5.284)
Statistical Analysis 1: Comparison: Stannous Fluoride; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.93, 95% CI 2-sided [2.844 to 5.012] — [estimate comment as in outcome 2, analysis 1]

11. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Restrictions (4 Item Total From Section 2 Questions 1 to 4) at Week 20
Description: as for outcome 7
Time Frame: At Baseline and Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a Scale
  At Baseline | 19.55 (5.088)
  At Week 20: number analyzed (Participants) | 66
  At Week 20 | 15.50 (6.422)
  Change from Baseline at Week 20: number analyzed (Participants) | 66
  Change from Baseline at Week 20 | -3.94 (5.865)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs. Week 20; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.15, 95% CI 2-sided [3.063 to 5.232] — [estimate comment as in outcome 2, analysis 1]

12. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Restrictions (4 Item Total From Section 2 Questions 1 to 4) at Week 24
Description: as for outcome 7
Time Frame: At Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a Scale
  At Baseline | 19.55 (5.088)
  At Week 24: number analyzed (Participants) | 66
  At Week 24 | 14.91 (6.738)
  Change from Baseline at Week 24: number analyzed (Participants) | 66
  Change from Baseline at Week 24 | -4.53 (5.717)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 24; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.74, 95% CI 2-sided [3.654 to 5.823] — [estimate comment as in outcome 2, analysis 1]

13. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Adaptation (12 Item Total From Section 2 Questions 5 to 16) at Week 4
Description: All participants scored first 4 questions present in Domain Adaptation of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6=Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Adaptation domain consisted of following questions Q5: I have to change the way I eat or drink certain things, Q6: I have to be careful how I breathe on a cold day, Q7: I have leave some cold foods/drinks to warm up before having them, Q8: I have to cool some foods/drinks down before I can have them, Q9: I have to cut up some fruits before eating, Q10: I have to wear scarf over my mouth on cold days, Q11: I have avoided very cold drinks/foods, Q12: I have avoided very hot drinks/foods, Q13: when eating some foods I have made sure they don't touch certain teeth, Q14: I have changed the way I brush, Q15: I bite some foods in small pieces, and Q16: there are other foods I have avoided.
Time Frame: At Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 53.12 (13.582)
  At Week 4: number analyzed (Participants) | 67
  At Week 4 | 51.42 (13.596)
  Change from Baseline at Week 4: number analyzed (Participants) | 67
  Change from Baseline at Week 4 | -1.46 (9.711)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 4; Test type: Other; p = 0.4185, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.11, 95% CI 2-sided [-1.592 to 3.821] — Difference is the baseline score minus other weeks score such that a positive difference favour to test dentifrice. Week 0 = Baseline

14. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Adaptation (12 Item Total From Section 2 Questions 5 to 16) at Week 8
Description: as for outcome 13
Time Frame: At Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 53.12 (13.582)
  At Week 8: number analyzed (Participants) | 69
  At Week 8 | 46.43 (16.453)
  Change from Baseline at Week 8: number analyzed (Participants) | 69
  Change from Baseline at Week 8 | -6.80 (12.678)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 8; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.08, 95% CI 2-sided [4.391 to 9.764] — [estimate comment as in outcome 2, analysis 1]

15. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Adaptation (12 Item Total From Section 2 Questions 5 to 16) at Week 12
Description: as for outcome 13
Time Frame: At Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 53.12 (13.582)
  At Week 12: number analyzed (Participants) | 70
  At Week 12 | 45.04 (16.985)
  Change from Baseline at Week 12: number analyzed (Participants) | 70
  Change from Baseline at Week 12 | -8.27 (14.998)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 12; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.35, 95% CI 2-sided [5.674 to 11.026] — Difference is the baseline score minus other weeks score such that a positive difference favour to test dentifrice. Week 0 = Baseline Valu

16. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Adaptation (12 Item Total From Section 2 Questions 5 to 16) at Week 16
Description: as for outcome 13
Time Frame: At Baseline and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a Scale
  At Baseline | 53.12 (13.582)
  At Week 16: number analyzed (Participants) | 66
  At Week 16 | 42.59 (16.966)
  Change from Baseline at Week 16: number analyzed (Participants) | 66
  Change from Baseline at Week 16 | -10.45 (15.037)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 16; Test type: Other — Week 0 Vs Week 16; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 10.43, 95% CI 2-sided [7.708 to 13.158] — [estimate comment as in outcome 2, analysis 1]

17. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Adaptation (12 Item Total From Section 2 Questions 5 to 16) at Week 20
Description: as for outcome 13
Time Frame: At Baseline and Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score ona scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score ona scale
  At Baseline | 53.12 (13.582)
  At Week 20: number analyzed (Participants) | 66
  At Week 20 | 41.89 (18.607)
  Change from Baseline at Week 20: number analyzed (Participants) | 66
  Change from Baseline at Week 20 | -11.48 (15.304)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 20; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 11.73, 95% CI 2-sided [9.008 to 14.459] — [estimate comment as in outcome 2, analysis 1]

18. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Adaptation (12 Item Total From Section 2 Questions 5 to 16) at Week 24
Description: as for outcome 13
Time Frame: At Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 53.12 (13.582)
  At Week 24: number analyzed (Participants) | 66
  At Week 24 | 41.67 (19.449)
  Change from Baseline at Week 24: number analyzed (Participants) | 66
  Change from Baseline at Week 24 | -11.71 (16.270)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 24; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 11.96, 95% CI 2-sided [9.235 to 14.686] — [estimate comment as in outcome 2, analysis 1]

19. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Social Impact (5 Item Total From Section 2 Questions 17 to 21) at Week 4
Description: All participants scored first 5 questions present in Domain Social Impact of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6=Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Social Impact domain consisted of following questions Q17: Because of sensations I take longer than others to finish meal, Q18: I have to be careful what I eat when I am with others because of sensation in my teeth, Q19: I hide the way I am eating with others because of sensations in my teeth, Q20: I am unable to fully take part in conversations because of sensations in my teeth., Q21: Going to dentist is hard for me because I know it is going to be painful as a result of sensations in my teeth.
Time Frame: At Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a Scale
  At Baseline | 17.99 (6.138)
  At Week 4: number analyzed (Participants) | 67
  At Week 4 | 17.30 (6.110)
  Change from Baseline at Week 4: number analyzed (Participants) | 67
  Change from Baseline at Week 4 | -0.57 (4.265)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 vs Week 4; Test type: Other; p = 0.3415, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [-0.604 to 1.738] — [estimate comment as in outcome 2, analysis 1]

20. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Social Impact (5 Item Total From Section 2 Questions 17 to 21) at Week 8
Description: as for outcome 19
Time Frame: At Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 17.99 (6.138)
  At Week 8: number analyzed (Participants) | 69
  At Week 8 | 16.32 (6.701)
  Change from Baseline at Week 8: number analyzed (Participants) | 69
  Change from Baseline at Week 8 | -1.67 (5.524)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 8; Test type: Other; p = 0.0029, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.77, 95% CI 2-sided [0.610 to 2.935] — [estimate comment as in outcome 13, analysis 1]

21. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Social Impact (5 Item Total From Section 2 Questions 17 to 21) at Week 12
Description: as for outcome 19
Time Frame: At Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 17.99 (6.138)
  At Week 12: number analyzed (Participants) | 70
  At Week 12 | 15.60 (6.787)
  Change from Baseline at Week 12: number analyzed (Participants) | 70
  Change from Baseline at Week 12 | -2.64 (6.459)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 12; Test type: Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.42, 95% CI 2-sided [1.266 to 3.582] — [estimate comment as in outcome 2, analysis 1]

22. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Social Impact (5 Item Total From Section 2 Questions 17 to 21) at Week 16
Description: as for outcome 19
Time Frame: At Baseline and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score ona Scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score ona Scale
  At Baseline | 17.99 (6.138)
  At Week 16: number analyzed (Participants) | 66
  At Week 16 | 14.44 (6.528)
  Change from Baseline at Week 16: number analyzed (Participants) | 66
  Change from Baseline at Week 16 | -3.62 (6.144)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 vs Week 16; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.55, 95% CI 2-sided [2.371 to 4.729] — [estimate comment as in outcome 2, analysis 1]

23. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Social Impact (5 Item Total From Section 2 Questions 17 to 21) at Week 20
Description: as for outcome 19
Time Frame: At Baseline and Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 17.99 (6.138)
  At Week 20: number analyzed (Participants) | 66
  At Week 20 | 13.79 (7.312)
  Change from Baseline at Week 20: number analyzed (Participants) | 66
  Change from Baseline at Week 20 | -4.33 (6.971)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 20; Test type: Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.39, 95% CI 2-sided [3.210 to 5.568] — [estimate comment as in outcome 2, analysis 1]

24. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Social Impact (5 Item Total From Section 2 Questions 17 to 21) at Week 24
Description: as for outcome 19
Time Frame: At Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 17.99 (6.138)
  At week 24: number analyzed (Participants) | 66
  At week 24 | 13.88 (7.154)
  Change from Baseline at Week 24: number analyzed (Participants) | 66
  Change from Baseline at Week 24 | -4.24 (6.730)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 24; Test type: Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.30, 95% CI 2-sided [3.119 to 5.477] — [estimate comment as in outcome 2, analysis 1]

25. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Emotional Impact (8 Item Total From Section 2 Questions 22 to 29) at Week 4
Description: All participants scored first 5 questions present in Domain Emotional Impact of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6=Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Emotional Impact domain consisted of following questions Q22: I've been frustrated because I can't find anything that deals with the sensations I have in my teeth. Q23: I have been anxious that something I eat or drink might cause sensations in my teeth, Q24: The sensations in my teeth have been irritating, Q25: I have been annoyed with myself because I did something that I knew caused these sensation, Q26: I felt guilty because I might have contributed to the sensations I am having with my teeth, Q27: the sensations in my teeth have been annoying, Q28: The sensations in my teeth have been embarrassing, Q29: I have been anxious because of the sensations in my teeth.
Time Frame: At Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a Scale
  At Baseline | 35.48 (9.106)
  At Week 4: number analyzed (Participants) | 67
  At Week 4 | 32.64 (8.388)
  Change from Baseline at Week 4: number analyzed (Participants) | 67
  Change from Baseline at Week 4 | -2.40 (6.649)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 4; Test type: Other; p = 0.0145, ANOVA; Mean Difference (Final Values) = 2.42, 95% CI 2-sided [0.483 to 4.352] — [estimate comment as in outcome 2, analysis 1]

26. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Emotional Impact (8 Item Total From Section 2 Questions 22 to 29) at Week 8
Description: as for outcome 25
Time Frame: At Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 35.48 (9.106)
  At Week 8: number analyzed (Participants) | 69
  At Week 8 | 31.42 (10.322)
  Change from Baseline at Week 8: number analyzed (Participants) | 69
  Change from Baseline at Week 8 | -4.30 (8.742)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 8; Test type: Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.42, 95% CI 2-sided [2.498 to 6.339] — [estimate comment as in outcome 2, analysis 1]

27. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Emotional Impact (8 Item Total From Section 2 Questions 22 to 29) at Week 12
Description: as for outcome 25
Time Frame: At Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a Scale
  At Baseline | 35.48 (9.106)
  At Week 12: number analyzed (Participants) | 70
  At Week 12 | 28.79 (11.518)
  Change from Baseline at Week 12: number analyzed (Participants) | 70
  Change from Baseline at Week 12 | -6.86 (11.119)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 12; Test type: Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.85, 95% CI 2-sided [4.933 to 8.759] — [estimate comment as in outcome 2, analysis 1]

28. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Emotional Impact (8 Item Total From Section 2 Questions 22 to 29) at Week 16
Description: as for outcome 25
Time Frame: At Baseline and Week 16
Population: The intention to treat (ITT) population was the primary population of analysis, defined as all participants who received the study toothpaste and had at least one post - baseline DHEQ/clinical assessm
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 35.48 (9.106)
  At Week 16: number analyzed (Participants) | 66
  At Week 16 | 28.24 (10.722)
  Change from Baseline at Week 16: number analyzed (Participants) | 66
  Change from Baseline at Week 16 | -7.33 (10.316)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 16; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.17, 95% CI 2-sided [5.219 to 9.115] — [estimate comment as in outcome 2, analysis 1]

29. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Emotional Impact (8 Item Total From Section 2 Questions 22 to 29) at Week 20
Description: as for outcome 25
Time Frame: At Baseline and Week 20
Population: The intention to treat (ITT) population was the primary population of analysis, defined as all participants who received the study toothpaste and had at least one post - baseline DHEQ/clinical assessme
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 35.48 (9.106)
  At week 20: number analyzed (Participants) | 66
  At week 20 | 27.32 (12.800)
  Change from Baseline at Week 20: number analyzed (Participants) | 66
  Change from Baseline at Week 20 | -8.17 (11.493)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 20; Test type: Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.39, 95% CI 2-sided [6.438 to 10.335] — [estimate comment as in outcome 2, analysis 1]

30. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Emotional Impact (8 Item Total From Section 2 Questions 22 to 29) at Week 24
Description: as for outcome 25
Time Frame: At Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 35.48 (9.106)
  At Week 24: number analyzed (Participants) | 66
  At Week 24 | 27.03 (12.701)
  Change from Baseline at Week 24: number analyzed (Participants) | 66
  Change from Baseline at Week 24 | -8.45 (12.158)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs. Week 24; Test type: Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.67, 95% CI 2-sided [6.726 to 10.623] — [estimate comment as in outcome 2, analysis 1]

31. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Identity (5 Item Total From Section 2 Questions 30 to 34) at Week 4
Description: All participants scored first 4 questions present in Domain Identity of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6=Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Identity domain consisted of following questions Q30: I find it difficult to accept that I am a person who has these sensations in my teeth, Q31: Having these sensations in my teeth makes me feel different from others, Q32:Having these sensations in my teeth makes me feel old, Q33:Having these sensations in my teeth makes me feel damaged, Q34: Having these sensations in my teeth makes me feel as though I am unhealthy.
Time Frame: At Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 16.27 (7.256)
  At Week 4: number analyzed (Participants) | 67
  At Week 4 | 15.66 (7.300)
  Change from Baseline at Week 4: number analyzed (Participants) | 67
  Change from Baseline at Week 4 | -0.64 (5.804)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 4; Test type: Other; p = 0.3676, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-0.738 to 1.989] — [estimate comment as in outcome 2, analysis 1]

32. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Identity (5 Item Total From Section 2 Questions 30 to 34) at Week 8
Description: as for outcome 31
Time Frame: At Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 16.27 (7.256)
  At Week 8: number analyzed (Participants) | 69
  At Week 8 | 15.55 (7.295)
  Change from Baseline at Week 8: number analyzed (Participants) | 69
  Change from Baseline at Week 8 | -0.81 (6.314)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 8; Test type: Other; p = 0.1907, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.90, 95% CI 2-sided [-0.451 to 2.255] — [estimate comment as in outcome 2, analysis 1]

33. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Identity (5 Item Total From Section 2 Questions 30 to 34) at Week 12
Description: All participants scored first 4 questions present in Domain Identity of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6=Agree, 5= Agree a little, 4= neither agree or disagree, 3= disagree a little, 2= disagree, and 1= strongly disagree. Restriction domain consisted of following questions Q30: I find it difficult to accept that I am a person who has these sensations in my teeth, Q31: Having these sensations in my teeth makes me feel different from others, Q32:Having these sensations in my teeth makes me feel old, Q33:Having these sensations in my teeth makes me feel damaged, Q34: Having these sensations in my teeth makes me feel as though I am unhealthy.
Time Frame: At Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 16.27 (7.256)
  At Week 12: number analyzed (Participants) | 70
  At Week 12 | 14.64 (7.404)
  Change from Baseline at Week 12: number analyzed (Participants) | 70
  Change from Baseline at Week 12 | -1.83 (7.305)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs. Week 12; Test type: Other; p = 0.0085, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.81, 95% CI 2-sided [0.467 to 3.162] — [estimate comment as in outcome 2, analysis 1]

34. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Identity (5 Item Total From Section 2 Questi 30 to 34) at Week 16
Description: All participants scored first 4 questions present in Domain Identity of section 2 of the DHEQ using a 7-point scale, where 7= Strongly agree, 6=Agree, 5= Agree a little, 4= neither agree or disagree, 3 disagree a little, 2= disagree, and 1= strongly disagree. Identity domain consisted of following questions Q30: I find it difficult to accept that I am a person who has these sensations in my teeth, Q31: Having these sensations in my teeth makes me feel different from others, Q32:Having these sensations in my teeth makes me feel old, Q33:Having these sensations in my teeth makes me fee damaged, Q34: Having these sensations in my teeth makes me feel as though I am unhealthy.
Time Frame: At Baseline and Week 16
Population: The intention to treat (ITT) population was the primary population of analysis, defined as all participants who received the study toothpa and had at least one post - baseline DHEQ/clinical assessment.
Measure: Mean (Standard Deviation); unit: Score ona scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score ona scale
  At Baseline | 16.27 (7.256)
  At Week 16: number analyzed (Participants) | 66
  At Week 16 | 14.55 (8.079)
  Change from Baseline at Week 16: number analyzed (Participants) | 66
  Change from Baseline at Week 16 | -2.29 (8.105)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 16; Test type: Other; p = 0.0026, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.12, 95% CI 2-sided [0.744 to 3.489] — [estimate comment as in outcome 2, analysis 1]

35. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Identity (5 Item Total From Section 2 Questions 30 to 34) at Week 20
Description: as for outcome 31
Time Frame: At Baseline and Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 16.27 (7.256)
  At Week 20: number analyzed (Participants) | 66
  At Week 20 | 13.82 (8.320)
  Change from Baseline at Week 20: number analyzed (Participants) | 66
  Change from Baseline at Week 20 | -2.65 (8.950)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 20; Test type: Other; p = 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.74, 95% CI 2-sided [1.371 to 4.116]

36. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Identity (5 Item Total From Section 2 Questions 30 to 34) at Week 24
Description: as for outcome 31
Time Frame: At Baseline and Week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 16.27 (7.256)
  At Week 24: number analyzed (Participants) | 66
  At Week 24 | 13.71 (8.364)
  Change from Baseline at Week 24: number analyzed (Participants) | 66
  Change from Baseline at Week 24 | -2.76 (8.769)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 vs Week 24; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.85, 95% CI 2-sided [1.477 to 4.222] — [estimate comment as in outcome 2, analysis 1]

37. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Global Oral Health Rating (Response to Section 2 Question 35) at Week 4
Description: All participants scored one question present in Domain Global oral health rating Global oral health rating of section 2 of the DHEQ using a 6-point scale, where, 6=Very poor, 5= poor, 4= Fair, 3= Good, 2=Very good, and 1= excellent. Global oral health rating domain consisted of following questionsQ35: overall how would you rate the health of your mouth, teeth and gums?
Time Frame: At Baseline and Week 4
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline: number analyzed (Participants) | 72
  At Baseline | 3.38 (0.926)
  At Week 4: number analyzed (Participants) | 67
  At Week 4 | 3.24 (0.889)
  Change from Baseline at Week 4: number analyzed (Participants) | 66
  Change from Baseline at Week 4 | -0.14 (0.654)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 4; Test type: Other; p = 0.2326, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.059 to 0.243] — [estimate comment as in outcome 15, analysis 1]

38. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Global Oral Health Rating (Response to Section 2 Question 35) at Week 8
Description: as for outcome 37
Time Frame: At Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline: number analyzed (Participants) | 72
  At Baseline | 3.38 (0.926)
  At Week 8: number analyzed (Participants) | 69
  At Week 8 | 3.32 (0.947)
  Change from Baseline at Week 8: number analyzed (Participants) | 68
  Change from Baseline at Week 8 | -0.04 (0.721)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 vs Week 8; Test type: Other; p = 0.3934, ANOVA — From ANOVA model with visit and site as fixed effect and subject as random effect. Visit*site interaction included where significant at 10% level; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.085 to 0.216] — [estimate comment as in outcome 2, analysis 1]

39. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Global Oral Health Rating (Response to Section 2 Question 35) at Week 12
Description: as for outcome 37
Time Frame: At Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline: number analyzed (Participants) | 72
  At Baseline | 3.38 (0.926)
  At Week 12: number analyzed (Participants) | 70
  At Week 12 | 3.27 (0.850)
  Change from Baseline at Week 12: number analyzed (Participants) | 69
  Change from Baseline at Week 12 | -0.12 (0.697)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 12; Test type: Other; p = 0.0795, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.016 to 0.284] — [estimate comment as in outcome 2, analysis 1]

40. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Global Oral Health Rating (Response to Section 2 Question 35) at Week 16
Description: All participants scored one question present in Domain Global oral health rating of section 2 of the DHEQ using a 6-point scale, where, 6=Very poor, 5= poor, 4= Fair, 3= Good, 2=Very good, and 1= excellent. Global oral health rating domain consisted of following questionsQ35: overall how would you rate the health of your mouth, teeth and gums?
Time Frame: At Baseline and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline: number analyzed (Participants) | 72
  At Baseline | 3.38 (0.92)
  At Week 16: number analyzed (Participants) | 66
  At Week 16 | 3.24 (0.912)
  Change from Baseline at Week 16: number analyzed (Participants) | 66
  Change from Baseline at Week 16 | -0.14 (0.788)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 vs Week 16; Test type: Other; p = 0.0682, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.011 to 0.294] — [estimate comment as in outcome 2, analysis 1]

41. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Global Oral Health Rating (Response to Section 2 Question 35) at Week 20
Description: as for outcome 40
Time Frame: At Baseline and Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline: number analyzed (Participants) | 72
  At Baseline | 3.38 (0.926)
  At Week 20: number analyzed (Participants) | 66
  At Week 20 | 3.29 (0.941)
  Change from Baseline at Week 20: number analyzed (Participants) | 65
  Change from Baseline at Week 20 | -0.11 (0.831)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 vs Week 20; Test type: Other; p = 0.0844, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.018 to 0.287] — [estimate comment as in outcome 2, analysis 1]

42. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Global Oral Health Rating (Response to Section 2 Question 35) at Week 24
Description: as for outcome 40
Time Frame: At Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline: number analyzed (Participants) | 72
  At Baseline | 3.38 (0.926)
  At Week 24: number analyzed (Participants) | 66
  At Week 24 | 3.24 (0.946)
  Change from Baseline at Week 24: number analyzed (Participants) | 65
  Change from Baseline at Week 24 | -0.15 (0.755)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 24; Test type: Other; p = 0.0211, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [0.027 to 0.332] — [estimate comment as in outcome 2, analysis 1]

43. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Effect on Life Overall (4 Item Total From Section 2 Questions 36 to 39) at Week 4
Description: All participants scored first 4 questions present in Domain Effect on Life Overall of section 2 of the DHEQ using a 5-point scale, 4= Very Much, 3= Quite a bit, 2= somewhat, and 1= a little, 0=not al all. Effect on Life Overall domain consisted of following questions Q36: Overall how much do the sensations in your teeth bother you? Q37: Overall, how much do the things you do to manage the sensations bother you? Q38: Overall, how much do the sensations in your teeth affect your quality of life? Q39: Overall, how much do the things you do to manage the sensations in your teeth affect your quality of life?
Time Frame: At Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 6.56 (3.539)
  At Week 4: number analyzed (Participants) | 67
  At Week 4 | 5.88 (3.278)
  Change from Baseline at Week 4: number analyzed (Participants) | 67
  Change from Baseline at Week 4 | -0.64 (2.515)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 vs Week 4; Test type: Other; p = 0.0493, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [0.002 to 1.194] — [estimate comment as in outcome 2, analysis 1]

44. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Effect on Life Overall (4 Item Total From Section 2 Questions 36 to 39) at Week 8
Description: as for outcome 43
Time Frame: At Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 6.56 (3.539)
  At Week 8: number analyzed (Participants) | 69
  At Week 8 | 5.12 (3.292)
  Change from Baseline at Week 8: number analyzed (Participants) | 69
  Change from Baseline at Week 8 | -1.43 (2.757)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 vs Week 8; Test type: Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.42, 95% CI 2-sided [0.830 to 2.013] — [estimate comment as in outcome 2, analysis 1]

45. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Effect on Life Overall (4 Item Total From Section 2 Questions 36 to 39) at Week 12
Description: : All participants scored first 4 questions present in Domain Effect on Life Overall of section 2 of the DHEQ using a 5-point scale, 4= Very Much, 3= Quite a bit, 2= somewhat, and 1= a little, 0=not al all. Effect on Life Overall domain consisted of following questions Q36: Overall how much do the sensations in your teeth bother you? Q37: Overall, how much do the things you do to manage the sensations bother you? Q38: Overall, how much do the sensations in your teeth affect your quality of life? Q39: Overall, how much do the things you do to manage the sensations in your teeth affect your quality of life?
Time Frame: At Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 6.56 (3.539)
  At Week 12: number analyzed (Participants) | 70
  At Week 12 | 4.70 (3.276)
  Change from Baseline at Week 12: number analyzed (Participants) | 70
  Change from Baseline at Week 12 | -1.87 (3.139)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 12; Test type: Other; p < 0.0001, ANOVA — [p-value comment as in outcome 38, analysis 1]; Mean Difference (Final Values) = 1.87, 95% CI 2-sided [1.278 to 2.457] — [estimate comment as in outcome 2, analysis 1]

46. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Effect on Life Overall (4 Item Total From Section 2 Questions 36 to 39) at Week 16
Description: as for outcome 43
Time Frame: At Baseline and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 6.56 (3.539)
  At Week 16: number analyzed (Participants) | 66
  At Week 16 | 4.42 (3.054)
  Change from Baseline at Week 16: number analyzed (Participants) | 66
  Change from Baseline at Week 16 | -2.12 (3.218)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 16; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.03, 95% CI 2-sided [1.429 to 2.629] — [estimate comment as in outcome 2, analysis 1]

47. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Effect on Life Overall (4 Item Total From Section 2 Questions 36 to 39) at Week 20
Description: as for outcome 43
Time Frame: At Baseline and Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 6.56 (3.539)
  At Week 20: number analyzed (Participants) | 66
  At Week 20 | 4.29 (3.436)
  Change from Baseline at Week 20: number analyzed (Participants) | 66
  Change from Baseline at Week 20 | -2.32 (3.613)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 20; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.34, 95% CI 2-sided [1.743 to 2.943] — [estimate comment as in outcome 2, analysis 1]

48. Primary Outcome: Change From Baseline in Mean DHEQ Score of Domain - Effect on Life Overall (4 Item Total From Section 2 Questions 36 to 39) at Week 24
Description: as for outcome 43
Time Frame: At Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 6.56 (3.539)
  At Week 24: number analyzed (Participants) | 66
  At Week 24 | 4.29 (3.281)
  Change from Baseline at Week 24: number analyzed (Participants) | 66
  Change from Baseline at Week 24 | -2.32 (3.407)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 24; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.34, 95% CI 2-sided [1.743 to 2.943] — [estimate comment as in outcome 2, analysis 1]

49. Primary Outcome: Change From Baseline in Mean Score of Dentine Hyersensitivity Experience Questionnaire (DHEQ) Section1 - Question (Q) No. 7 At Week 4
Description: All the participants scored question No. 7 (Q7: on a scale of 1 to 10 how intense are the sensations?) of section 1 of DHEQ on a scale of 1 to 10, where 1 =not at all intense and 10= worst imaginable. Section 1 of DHEQ consisted questions about participant's sensitive teeth and the impact they had on participant's everyday life.
Time Frame: At Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 5.78 (1.677)
  At Week 4: number analyzed (Participants) | 67
  At Week 4 | 4.85 (1.598)
  Change from Baseline at Week 4: number analyzed (Participants) | 67
  Change from Baseline at Week 4 | -0.88 (1.805)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 4; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.88, 95% CI 2-sided [0.474 to 1.295] — [estimate comment as in outcome 2, analysis 1]

50. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 7 At Week 8
Description: as for outcome 49
Time Frame: At Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 5.78 (1.677)
  At Week 8: number analyzed (Participants) | 69
  At Week 8 | 4.49 (1.720)
  Change from Baseline at Week 8: number analyzed (Participants) | 69
  Change from Baseline at Week 8 | -1.26 (1.968)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 8; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.28, 95% CI 2-sided [0.875 to 1.690] — [estimate comment as in outcome 2, analysis 1]

51. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 7 At Week 12
Description: as for outcome 49
Time Frame: At Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 5.78 (1.677)
  At Week 12: number analyzed (Participants) | 70
  At Week 12 | 4.01 (1.830)
  Change from Baseline at Week 12: number analyzed (Participants) | 70
  Change from Baseline at Week 12 | -1.73 (2.139)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 12; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.74, 95% CI 2-sided [1.333 to 2.145] — [estimate comment as in outcome 2, analysis 1]

52. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 7 At Week 16
Description: as for outcome 49
Time Frame: At Baseline and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 5.78 (1.677)
  At Week 16: number analyzed (Participants) | 66
  At Week 16 | 3.74 (1.809)
  Change from Baseline at Week 16: number analyzed (Participants) | 66
  Change from Baseline at Week 16 | -1.98 (2.042)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 16; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.96, 95% CI 2-sided [1.545 to 2.371] — [estimate comment as in outcome 2, analysis 1]

53. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 7 At Week 20
Description: as for outcome 49
Time Frame: At Baseline and Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 5.78 (1.677)
  At Week 20: number analyzed (Participants) | 66
  At Week 20 | 3.67 (1.940)
  Change from Baseline at Week 20: number analyzed (Participants) | 66
  Change from Baseline at Week 20 | -2.06 (2.045)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs. Week 20; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.06, 95% CI 2-sided [1.643 to 2.469] — [estimate comment as in outcome 2, analysis 1]

54. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 7 At Week 24
Description: as for outcome 49
Time Frame: At Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 5.78 (1.677)
  At Week 24: number analyzed (Participants) | 66
  At Week 24 | 3.52 (1.791)
  Change from Baseline at Week 24: number analyzed (Participants) | 66
  Change from Baseline at Week 24 | -2.21 (2.116)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 24; Test type: Other; p < .0001, ANOVA — [p-value comment as in outcome 38, analysis 1]; Mean Difference (Final Values) = 2.21, 95% CI 2-sided [1.794 to 2.620] — [estimate comment as in outcome 2, analysis 1]

55. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 8 At Week 4
Description: All the participants scored question No. 8 (Q8: on a scale of 1 to 10 how bothered are you by any sensations?) of section 1 of DHEQ on a scale of 1 to 10, where 1 =not at all bothered and 10= extremely bothered. Section 1 of DHEQ consisted questions about participant's sensitive teeth and the impact they had on participant's everyday life.
Time Frame: At Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 5.93 (2.226)
  At Week 4: number analyzed (Participants) | 67
  At Week 4 | 4.69 (1.924)
  Change from Baseline at Week 4: number analyzed (Participants) | 67
  Change from Baseline at Week 4 | -1.22 (2.014)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 4; Test type: Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.18, 95% CI 2-sided [0.703 to 1.660] — [estimate comment as in outcome 2, analysis 1]

56. Primary Outcome: Change From Baseline in Mean Score DHEQ Section1 - Question (Q) No. 8 At Week 8
Description: as for outcome 55
Time Frame: At Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 5.93 (2.226)
  At Week 8: number analyzed (Participants) | 69
  At Week 8 | 4.51 (1.960)
  Change from Baseline at Week 8: number analyzed (Participants) | 69
  Change from Baseline at Week 8 | -1.45 (2.304)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 8; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.45, 95% CI 2-sided [0.977 to 1.926] — [estimate comment as in outcome 2, analysis 1]

57. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 8 At Week 12
Description: All the participants scored question No. 8 (Q8: on a scale of 1 to 10 how bothered are you by any sensations?) of section 1 of DHEQ on a scale of 1 to 10, where 1 =not at all bothered and 10= extremely bothered. Section 1 of DHEQ consisted questions about participant's sensitive teeth and impact they had on participant's everyday life.
Time Frame: At Baseline and Week 12
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 5.93 (2.226)
  At Week 12: number analyzed (Participants) | 70
  At Week 12 | 3.99 (2.054)
  Change from Baseline at Week 12: number analyzed (Participants) | 70
  Change from Baseline at Week 12 | -1.94 (2.670)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 12; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.95, 95% CI 2-sided [1.473 to 2.418] — [estimate comment as in outcome 2, analysis 1]

58. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 8 At Week 16
Description: as for outcome 55
Time Frame: At Baseline and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 5.93 (2.226)
  At Week 16: number analyzed (Participants) | 66
  At Week 16 | 3.55 (1.773)
  Change from Baseline at Week 16: number analyzed (Participants) | 66
  Change from Baseline at Week 16 | -2.35 (2.657)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week16; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.33, 95% CI 2-sided [1.848 to 2.810] — [estimate comment as in outcome 2, analysis 1]

59. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 8 At Week20
Description: as for outcome 55
Time Frame: At Baseline and Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 5.93 (2.226)
  At Week 20: number analyzed (Participants) | 66
  At Week 20 | 3.70 (2.068)
  Change from Baseline at Week 20: number analyzed (Participants) | 66
  Change from Baseline at Week 20 | -2.20 (2.591)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs. Week 20; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.21, 95% CI 2-sided [1.732 to 2.694] — [estimate comment as in outcome 2, analysis 1]

60. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 8 At Week 24
Description: as for outcome 55
Time Frame: At Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a Scale
  At Baseline | 5.93 (2.226)
  At Week 24: number analyzed (Participants) | 66
  At Week 24 | 3.41 (1.848)
  Change from Baseline at Week 24: number analyzed (Participants) | 66
  Change from Baseline at Week 24 | -2.48 (2.562)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 Vs Week 24; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.50, 95% CI 2-sided [2.020 to 2.982] — [estimate comment as in outcome 2, analysis 1]

61. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 9 At Week 4
Description: All the participants scored question No. 9 (Q9: on a scale of 1 to 10 how well can you tolerate sensations?) of section 1 of DHEQ on a scale of 1 to 10, where 1 =can easily tolerate and 10= cannot tolerate at all. Section 1 of DHEQ consisted questions about participant's sensitive teeth and the impact they had on participant's everyday life.
Time Frame: At Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 4.95 (2.040)
  At Week 4: number analyzed (Participants) | 67
  At Week 4 | 4.46 (1.861)
  Change from Baseline at Week 4: number analyzed (Participants) | 67
  Change from Baseline at Week 4 | -0.43 (1.885)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 vs Week 4; Test type: Other; p = 0.0786, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-0.050 to 0.919] — [estimate comment as in outcome 2, analysis 1]

62. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 9 at Week 8
Description: as for outcome 61
Time Frame: At Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 4.95 (2.040)
  At Week 8: number analyzed (Participants) | 69
  At Week 8 | 4.29 (2.087)
  Change from Baseline at Week 8: number analyzed (Participants) | 69
  Change from Baseline at Week 8 | -0.67 (2.501)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 vs Week 8; Test type: Other; p = 0.0050, ANOVA; [1] From ANOVA model with visit and site as fixed effect and subject as random effect. Visit*site interaction included where significant at 10% level; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [0.210 to 1.171] — [estimate comment as in outcome 2, analysis 1]

63. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 9 At Week 12
Description: as for outcome 61
Time Frame: At Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 4.95 (2.040)
  At Week 12: number analyzed (Participants) | 70
  At Week 12 | 3.56 (1.878)
  Change from Baseline at Week 12: number analyzed (Participants) | 70
  Change from Baseline at Week 12 | -1.39 (2.373)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 vs Week 12; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.40, 95% CI 2-sided [0.918 to 1.875] — [estimate comment as in outcome 2, analysis 1]

64. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 9 At Week 16
Description: as for outcome 61
Time Frame: At Baseline and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 4.95 (2.040)
  At Week 16: number analyzed (Participants) | 66
  At Week 16 | 3.47 (1.684)
  Change from baseline at Week 16: number analyzed (Participants) | 66
  Change from baseline at Week 16 | -1.47 (2.374)
Statistical Analysis 1: Comparison: Stannous Fluoride; Test type: Other; p < .0001, ANOVA; [From ANOVA model with visit and site as fixed effect and subject as random effect. Visit*site interaction included where significant at 10% level; Mean Difference (Final Values) = 1.44, 95% CI 2-sided [0.951 to 1.926] — [estimate comment as in outcome 2, analysis 1]

65. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 9 At Week 20
Description: as for outcome 61
Time Frame: At Baseline and Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 4.95 (2.040)
  At Week 20: number analyzed (Participants) | 66
  At Week 20 | 3.76 (2.134)
  Change from Baseline at Week 20: number analyzed (Participants) | 66
  Change from Baseline at Week 20 | -1.17 (2.415)
Statistical Analysis 1: Comparison: Stannous Fluoride; Week 0 vs Week 20; Test type: Other; p < .0001, ANOVA — [p-value comment as in outcome 38, analysis 1]; Mean Difference (Final Values) = 1.17, 95% CI 2-sided [0.678 to 1.653] — [estimate comment as in outcome 2, analysis 1]

66. Primary Outcome: Change From Baseline in Mean Score of DHEQ Section1 - Question (Q) No. 9 At Week 24
Description: as for outcome 61
Time Frame: At Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride
Number analyzed (Participants) | 73
Score on a scale
  At Baseline | 4.95 (2.040)
  At Week 24: number analyzed (Participants) | 66
  At Week 24 | 3.36 (1.911)
  Change from baseline at Week 24: number analyzed (Participants) | 66
  Change from baseline at Week 24 | -1.56 (2.620)
Statistical Analysis 1: Comparison: Stannous Fluoride; Test type: Other; p < .0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.56, 95% CI 2-sided [1.072 to 2.047] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline to Week 24
Groups:
- Stannous Fluoride: Participants will brush with a full brush head of toothpaste for 1 timed minute (in their usual manner), twice daily (morning and evening) from baseline
Arm/Group | Stannous Fluoride
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 1/75
Other Adverse Events (participants affected / at risk) | 47/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stannous Fluoride (N=75)
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stannous Fluoride (N=75)
ORAL HERPES (Infections and infestations) | 12
ORAL HERPES (Infections and infestations) | 7
GASTROENTERITIS (Infections and infestations) | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3
HERPES VIRUS INFECTION (Infections and infestations) | 1
OTITIS MEDIA (Infections and infestations) | 1
TONSILLITIS BACTERIAL (Infections and infestations) | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
PHARYNGITIS (Infections and infestations) | 1
CONJUNCTIVITIS (Infections and infestations) | 1
TOOTHACHE (Gastrointestinal disorders) | 5
ORAL MUCOSAL EXFOLIATION (Gastrointestinal disorders) | 4
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
GINGIVAL BLEEDING (Gastrointestinal disorders) | 21
LIP EXFOLIATION (Gastrointestinal disorders) | 1
LIP ULCERATION (Gastrointestinal disorders) | 2
MOUTH ULCERATION (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
ORAL MUCOSAL ERYTHEMA (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 2
APHTHOUS ULCER (Gastrointestinal disorders) | 1
ORAL DISCOMFORT (Gastrointestinal disorders) | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 3
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 3
TOOTH INJURY (Injury, poisoning and procedural complications) | 2
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1
EYELID INJURY (Injury, poisoning and procedural complications) | 1
FACE INJURY (Injury, poisoning and procedural complications) | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 1
POST-TRAUMATIC NECK SYNDROME (Injury, poisoning and procedural complications) | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1
TRAUMATIC ULCER (Injury, poisoning and procedural complications) | 1
MOUTH INJURY (Injury, poisoning and procedural complications) | 1
HEADACHE (Nervous system disorders) | 12
DEVICE FAILURE (Product Issues) | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2
EAR PAIN (Ear and labyrinth disorders) | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT02752958/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT02752958/SAP_001.pdf